CLINICAL TRIAL: NCT05654116
Title: The Copenhagen Daycare Project: Enhancing the Role of Daycare Providers in Supporting Young Children's Social and Emotional Development
Brief Title: Testing the Effects of the Caregiver Interaction Profile Training on the Interactive Skills of Daycare Providers
Acronym: CDP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Copenhagen (Other)
Collaborators: Copenhagen Municipality, Denmark (Other Government); University College Copenhagen (Other); University of Groningen (Other); VU University of Amsterdam (Other)
Responsible Party: Principal Investigator, Sophie Reijman, Assistant professor, University of Copenhagen
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 514-0217/21-2000
Record Dates: First submitted 2022-12-01; First posted 2022-12-16 (Actual); Last update posted 2024-01-05 (Actual); Status verified 2024-01

CONDITIONS: Healthy; Emotion Regulation; Language Development; Interactive Skills Daycare Providers
MeSH Terms: conditions — Emotional Regulation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Trained coders who code the outcome variables of the study (from video-recorded material) will be blind to the intervention vs control condition, and to the baseline vs follow-up condition.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CIP training group (Experimental): Participants assigned to the CIP training group will receive either an individual 5-week CIP training or a pairwise 6-week CIP training, both with weekly sessions.
  Interventions: Behavioral: Caregiver Interaction Profile (CIP) training
- Waiting-list control group (No Intervention): Participants assigned to the waiting-list control group will receive no intervention while data collection is ongoing; after data collection is finished they will also receive the CIP training.

INTERVENTIONS:
Behavioral: Caregiver Interaction Profile (CIP) training — The CIP training aims to boost six interactive skills in daycare providers: sensitive responsiveness, respect for children's autonomy, structuring and limit setting, verbal communication, developmental stimulation, and fostering positive peer interactions. The training takes place with 1 or 2 daycare providers at a time, and consists of 5 or 6 weekly sessions, respectively. In individual trainings, sessions 1-3 focus on two skills each, session 4 is a recap of two skills the daycare provider chooses, and the final session is shared with a colleague. In pairwise sessions, session 1 focuses on the first two skills, sessions 2-5 each focus on one skill, and the last session serves as a recap of two skills the daycare providers choose. The training uses a video-feedback method: daycare providers are filmed in interactions with children in daycare, the CIP trainer preselects relevant fragments of video recordings to discuss with the daycare provider(s) during the training sessions.
  Arms: CIP training group

SUMMARY:
The goal of this clinical trial is to test the Caregiver Interaction Profile (CIP) training program (Helmerhorst et al., 2017) promoting the relational quality between professional caregivers and children in daycare. The main questions it aims to answer are:

* Does the CIP training program, compared to no training, improve the relational quality between daycare providers and children in daycare?
* Does the CIP training program, compared to no training, foster children's social, emotional, and language development? Daycare providers assigned to the "training group" will participate in the CIP training program, which uses video-recorded interactions between the daycare providers and children in daycare to give feedback on the relational quality as observed in the videos. Daycare providers assigned to the "waiting list control group" will initially not take part in the training program but will receive the training after the study is finished. All daycare providers' daily interactions with the children in daycare will be filmed before and after the training in order to see if there has been a change in relational quality for the daycare providers in the training group (compared to the control group). Daycare providers in the training and control groups will also fill out questionnaires about the social, emotional, and language development of the children in their care.

Researchers will compare daycare providers (and the children in their care) in the "training group" to daycare providers (and the children in their care) in the "control group" to see if the relational quality in the training group improves more than that in the control group as a result of the CIP training, and how that impacts the social, emotional, and language development of children.

ELIGIBILITY:
Inclusion Criteria:

* currently working as a professional daycare provider in a daycare center

Exclusion Criteria:

* temporary staff in daycare on short-term contracts

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2021-08-01 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Post-Training Scores on CIP Scale Sensitive Responsiveness | 9 weeks time frame between pre-training and post-training measurements for individual trainings; 10 weeks between pre-training and post-training measurements for pairwise trainings
  The degree to which daycare providers respond promptly and appropriately to children's signals, coded using the Caregiver Interaction Profile scales (Helmerhorst et al., 2014), rated from 1 (low) to 7 (high).
Post-Training Scores on CIP Scale Respect for Children's Autonomy | 9 weeks time frame between pre-training and post-training measurements for individual trainings; 10 weeks between pre-training and post-training measurements for pairwise trainings
  The degree to which daycare providers are not intrusive but validate and encourage children's ideas, initiatives and intentions, coded using the Caregiver Interaction Profile scales (Helmerhorst et al., 2014), rated from 1 (low) to 7 (high).
Post-Training Scores on CIP Scale Structuring and Limit Setting | 9 weeks time frame between pre-training and post-training measurements for individual trainings; 10 weeks between pre-training and post-training measurements for pairwise trainings
  The degree to which daycare providers structure activities in a way that children can benefit, and communicate clearly to children what is expected of them and ensure they comply with the expectations, coded using the Caregiver Interaction Profile scales (Helmerhorst et al., 2014), rated from 1 (low) to 7 (high).
Post-Training Scores on CIP Scale Verbal Communication | 9 weeks time frame between pre-training and post-training measurements for individual trainings; 10 weeks between pre-training and post-training measurements for pairwise trainings
  The degree to which daycare providers verbally interact with children, and the quality of their interactions (incl form, tone, content), coded using the Caregiver Interaction Profile scales (Helmerhorst et al., 2014), rated from 1 (low) to 7 (high).
Post-Training Scores on CIP Scale Developmental Stimulation | 9 weeks time frame between pre-training and post-training measurements for individual trainings; 10 weeks between pre-training and post-training measurements for pairwise trainings
  The degree to which daycare providers stimulate children's personal competencies (incl cognitive, creative, motor development), coded using the Caregiver Interaction Profile scales (Helmerhorst et al., 2014), rated from 1 (low) to 7 (high).
Post-Training Scores on CIP Scale Fostering Positive Peer Interactions | 9 weeks time frame between pre-training and post-training measurements for individual trainings; 10 weeks between pre-training and post-training measurements for pairwise trainings
  The degree to which daycare providers facilitate and stimulate children interacting with each other in positive ways, such as helping, comforting, sharing, collaborating, coded using the Caregiver Interaction Profile scales (Helmerhorst et al., 2014), rated from 1 (low) to 7 (high).

SECONDARY OUTCOMES:
Post-Training Scores on Ages and Stages Questionnaire: Social-Emotional, Daycare Provider-Report | 21 weeks time frame between pre-training and post-training assessments for individual trainings; 22 weeks time frame between pre-training and post-training assessments for pairwise trainings
  The Ages and Stages Questionnaire: Social-Emotional (ASQ:SE; Squires et al., 2001) measures signs of disturbances in children's socio-emotional development; higher scores reflect more indications of socio-emotional disturbances in development. The ASQ:SE is filled out by children's daycare providers. Items describe socio-emotional behaviours, and daycare providers indicate whether these apply "most of the time", "sometimes", or "rarely or never". They can check the item if it presents a particular concern for them, which increases the overall score.
Post-Training Scores on Ages and Stages Questionnaire: Social-Emotional, Parent-Report | 21 weeks time frame between pre-training and post-training assessments for individual trainings; 22 weeks time frame between pre-training and post-training assessments for pairwise trainings
  The Ages and Stages Questionnaire: Social-Emotional (ASQ:SE; Squires et al., 2001) measures signs of disturbances in children's socio-emotional development; higher scores reflect more indications of socio-emotional disturbances in development. The questionnaires are filled out by one of the children's parents. Items describe socio-emotional behaviours, and parents indicate whether these apply "most of the time", "sometimes", or "rarely or never". They can check the item if it presents a particular concern for them, which increases the overall score.
Post-Training Scores on Strengths and Difficulties Questionnaire, Daycare Provider-Report | 21 weeks time frame between pre-training and post-training assessments for individual trainings; 22 weeks time frame between pre-training and post-training assessments for pairwise trainings
  The Strengths and Difficulties Questionnaire (SDQ; Goodman, 2001) has 25 items about positive and negative attributes in children, such as how children behave in social relationships. Daycare providers indicate for each item on a 3-point scale to what degree it applies to the child in question. A total difficulties score is calculated, and a prosocial behavour (strength) score.
Post-Training Scores on Strengths and Difficulties Questionnaire, Parent-Report | 21 weeks time frame between pre-training and post-training assessments for individual trainings; 22 weeks time frame between pre-training and post-training assessments for pairwise trainings
  The Strengths and Difficulties Questionnaire (SDQ; Goodman, 2001) has 25 items about positive and negative attributes in children, such as how children behave in social relationships. Parents indicate for each item on a 3-point scale to what degree it applies to their child. A total difficulties score is calculated, and a prosocial behavour (strength) score.
Post-Training Scores on Child Behavior Checklist 1.5-5, Daycare Provider-Report | 21 weeks time frame between pre-training and post-training assessments for individual trainings; 22 weeks time frame between pre-training and post-training assessments for pairwise trainings
  The Child Behaviour Checklist 1.5-5 (CBCL 1.5-5; Achenbach & Rescorla, 2000) has 99 items measuring problem behavior in young children (such as "afraid to try new things"), with answer options "not true", "somewhat/sometimes true", and "very/often true". This questionnaire is filled out by daycare providers. Higher scores indicate higher levels of problem behavior.
Post-Training Scores on Child Behavior Checklist 1.5-5, Parent-Report | 21 weeks time frame between pre-training and post-training assessments for individual trainings; 22 weeks time frame between pre-training and post-training assessments for pairwise trainings
  The Child Behavior Checklist 1.5-5 (CBCL 1.5-5; Achenbach & Rescorla, 2000) has 99 items measuring problem behavior in young children (such as "afraid to try new things"), with answer options "not true", "somewhat/sometimes true", and "very/often true". This questionnaire is filled out by parents. Higher scores indicate higher levels of problem behavior.
Post-Training Scores on MacArthur Communicative Development Inventory-Short Form, Daycare Provider-Report | 21 weeks time frame between pre-training and post-training assessments for individual trainings; 22 weeks time frame between pre-training and post-training assessments for pairwise trainings
  The MacArthur Communicative Development Inventory-short, adapted for daycare (CDI-short; Bleses et al., 2018) has 70 vocabulary items, including animal sounds, body parts, and food and drink, which are checked by the daycare provider if they have heard the child produce the item, independent of pronunciation. More checks indicate more advanced communicative development.
Post-Training Scores on MacArthur Communicative Development Inventory-Short Form, Parent-Report | 21 weeks time frame between pre-training and post-training assessments for individual trainings; 22 weeks time frame between pre-training and post-training assessments for pairwise trainings
  The MacArthur Communicative Development Inventory-short, adapted for daycare (CDI-short; Bleses et al., 2018) has 70 vocabulary items, including animal sounds, body parts, and food and drink, which are checked by parents if they have heard their child produce the item, independent of pronunciation. More checks indicate more advanced communicative development.

CONTACTS AND LOCATIONS:
Overall Officials: Sophie Reijman, PhD, Principal Investigator — University of Copenhagen
Locations (1):
- Department of Psychology, University of Copenhagen, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Helmerhorst KOW, Riksen-Walraven JMA, Fukkink RG, Tavecchio LWC, Gevers Deynoot-Schaub MJJM. Effects of the Caregiver Interaction Profile Training on Caregiver-Child Interactions in Dutch Child Care Centers: A Randomized Controlled Trial. Child Youth Care Forum. 2017;46(3):413-436. doi: 10.1007/s10566-016-9383-9. Epub 2016 Nov 30. PMID 28490857
- [Background] Squires J, Bricker D, Heo K, Twombly E. Identification of social-emotional problems in young children using a parent-completed screening measure. Early Childhood Research Quarterly. 2001; 16(4): 405-419.
- [Background] Achenbach TM, Rescorla LA. Manual for the ASEBA Preschool Forms and Profiles. Burlington: University of Vermont, Research Center for Children, Youth, and Families; 2000.
- [Background] Goodman R. Psychometric properties of the strengths and difficulties questionnaire. J Am Acad Child Adolesc Psychiatry. 2001 Nov;40(11):1337-45. doi: 10.1097/00004583-200111000-00015. PMID 11699809
- [Background] Bleses D, Jensen P, Hojen A, Dale PS. An educator-administered measure of language development in young children. Infant Behav Dev. 2018 Aug;52:104-113. doi: 10.1016/j.infbeh.2018.06.002. Epub 2018 Jul 7. PMID 29990685
- [Background] Helmerhorst KOW, Riksen-Walraven JMA, Vermeer HJ, Fukkink RG, Tavecchio LWC. Measuring interactive skills of caregivers in child care centers: Development and validation of the caregiver interaction profile scales. Early Education and Development. 2014; 25(5): 770-790
- [Derived] Reijman S, Christensen Vieira C, Wahl Haase T, Helmerhorst KOW, Pontoppidan M, Grosen SA, Egmose I, Rohder K, Skovgaard Vaever M. A randomized trial of the Caregiver Interaction Profile (CIP) training with childcare providers: the Copenhagen Daycare Project study protocol. BMC Psychol. 2024 Mar 6;12(1):127. doi: 10.1186/s40359-024-01568-1. PMID 38449031